CLINICAL TRIAL: NCT01054937
Title: First-in-Man, Randomised, Double-Blind, Placebo-Controlled, Single Dose Escalation Study of the Novel Compound 4SC-203 in Young Healthy Volunteers
Brief Title: Single Dose Study With 4SC-203 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4SC AG (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4SC-203-2-2009
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: 4SC-203; Phase I; single dose; healthy volunteers
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 4SC-203 (Experimental)
  Interventions: Drug: 4SC-203
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4SC-203 — i.v. administration
  Arms: 4SC-203
Drug: Placebo — i.v. administration
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate safety and tolerability of 4SC-203 after a single dose administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years (included), and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening
* Subjects must be able to communicate well with the investigator, to understand and comply with the requirements of the study, and to understand and sign the written informed consent

Exclusion Criteria:

* Evidence of current or previous clinically significant disease, medical condition or finding of the medical examination (including vital signs and ECG), that in the opinion of the investigator would compromise the safety of the subject or the quality of the data
* Current or recent history of significant renal, hepatic, haematological, immunological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the subject's participation in the trial

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Investigation of safety and tolerability of escalating single doses of 4SC-203. | 14 days

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of single doses of 4SC-203. | 14 days
To assess the pharmacodynamic effect by means of appropriate biomarkers. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Frank Wagner, PD Dr. med., Principal Investigator — Charité Research Organisation GmbH, Berlin, Germany
Locations (1):
- Charité Research Organisation, Berlin, Germany